CLINICAL TRIAL: NCT06998784
Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Acute Pancreatitis: A Randomized Controlled Trial
Brief Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20242424
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-05

CONDITIONS: Acute Pancreatitis (AP); Vagus Nerve Stimulations
Keywords: acute pancreatitis; vagus nerve stimulations; PAN-PROMISE
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients will receive taVNS at left tragus up to 7 days.
  Interventions: Device: taVNS
- Sham-treatment group (Sham Comparator): Patients will receive sham-taVNS at left earlobe up to 7 days.
  Interventions: Device: Sham-taVNS

INTERVENTIONS:
Device: taVNS — Patients will receive taVNS at left tragus (a device developed by the Engineering Research Center of Molecular and Neuro Imaging, Ministry of Education (School of Life Science and Technology, Xidian University), in collaboration with the Wearable BCI and Intelligent Rehabilitation Innovation Lab (Guangzhou Institute of Technology, Xidian University)) twice daily (morning and night) for 30 minutes per session over a period of up to 7 days. The stimulation parameters are as follows:
  * Duty circle: 30s "on" periods alternating with 30s "off" periods;
  * Frequency: 25 Hz;
  * Amplitude: 0-2 mA (adjusted to the maximum tolerated level for each patient);
  * Pulse width: 0.5 ms.
  Arms: Treatment group
Device: Sham-taVNS — Patients will receive taVNS at left earlobe (a device developed by the Engineering Research Center of Molecular and Neuro Imaging, Ministry of Education (School of Life Science and Technology, Xidian University), in collaboration with the Wearable BCI and Intelligent Rehabilitation Innovation Lab (Guangzhou Institute of Technology, Xidian University)) twice daily (morning and night) for 30 minutes per session over a period of up to 7 days. The stimulation parameters are as follows: *Duty circle: 30s "on" periods alternating with 30s "off" periods; *Frequency: 25 Hz; *Amplitude: 0-2 mA (adjusted to the maximum tolerated level for each patient); *Pulse width: 0.5 ms.
  Arms: Sham-treatment group

SUMMARY:
Acute pancreatitis (AP), characterized by the sudden onset of pancreatic inflammation, is a frequent gastrointestinal emergency. Early suppression of the inflammatory response is critical to mitigate disease progression. When localized pancreatic inflammation progresses to systemic inflammation, triggering systemic inflammatory response syndrome (SIRS), the condition advances to moderate or severe AP, with mortality rates ranging from 10% to 40%. Additionally, early resumption of enteral nutrition reduces the risk of intra-abdominal infections and organ failure associated with AP. However, gastrointestinal dysfunction, which frequently manifests as gastroparesis or intestinal obstruction in severe cases , significantly complicates AP management by prolonging recovery time and compromising nutritional tolerance. Current early-phase management of AP remains suboptimal: anti-inflammatory strategies are predominantly limited to fluid resuscitation, while gastrointestinal function preservation is frequently underestimated. Consequently, effective therapies targeting both inflammatory suppression and gastrointestinal functional restoration in the early phase of AP are urgently needed.

The central nervous system plays a pivotal role in regulating peripheral immune responses, with the vagal anti-inflammatory signaling pathway serving as a key efferent pathway of the inflammatory reflex. Animal studies have shown a protective effect of the vagal anti-inflammatory signaling pathway against AP. Specifically, vagus nerve stimulation (VNS) significantly reduced pancreatic injury and improved survival in mice with severe AP. Furthermore, VNS has shown therapeutic potential in animal models of sepsis, shock, and renal ischemia-reperfusion injury, conditions frequently associated with systemic inflammation in severe pancreatitis. These findings suggest that VNS may alleviate both local and systemic inflammatory responses, as well as their complications.

Notably, prior clinical trial revealed that transcutaneous auricular VNS (taVNS) alleviated functional dyspepsia symptoms in adults, indicating its dual capacity for anti-inflammatory effects and gastrointestinal functional modulation. Based on this evidence, the investigators propose a randomized, sham-controlled trial to systematically evaluate the therapeutic efficacy of taVNS in patients with acute pancreatitis .

ELIGIBILITY:
Inclusion Criteria:

1. AP patients aged 18-80 years.
2. PAN-PROMISE score ≥15 and no participation in any other clinical trials within the past 3 months.

Exclusion Criteria:

1. Presence of diseases or conditions different from AP that may interfere with the scale, for example, other causes of abdominal pain (especially acute cholecystitis), obstruction of the digestive tract (peptic pyloric stenosis, gastrointestinal anastomotic stenosis, diabetic gastroparesis, gastrointestinal neoplasia...), nausea-vomiting (brain tumour, chemotherapy...) or weakness (pre-existing anaemia with haemoglobin <9 g/dL, heart failure or respiratory insufficiency associated with minimal effort dyspnoea, or domiciliary treatment with O2, advanced neoplasms or other debilitating diseases);
2. Implanted cardiac pacemaker or other electronic devices;
3. Prior treatment with transcutaneous auricular vagus nerve stimulation (taVNS);
4. Known malignancy;
5. Severe cardiovascular/cerebrovascular, hepatic, or renal diseases;
6. Cognitive impairment, psychiatric disorders, or other conditions that may affect patient cooperation;
7. Refusal to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Median treatment duration | Up to one week
  The number of treatment days required to reduce the PAN-PROMISE scores to 6. The PAN-PROMISE score (PAtieNt-rePoRted OutcoMe scale in acute pancreatItis from an international proSpEctive cohort study) consists of a seven-item scale based on the symptoms that cause the most discomfort and concern to patients with AP. Each symptom is rated on a scale of 0 to 10 points, where higher scores reflect greater symptom severity.

SECONDARY OUTCOMES:
PAN-PROMISE score during the study period | 1 week
  Change from baseline in PAN-PROMISE score during the study period.The PAN-PROMISE score (PAtieNt-rePoRted OutcoMe scale in acute pancreatItis from an international proSpEctive cohort study) consists of a seven-item scale based on the symptoms that cause the most discomfort and concern to patients with AP. Each symptom is rated on a scale of 0 to 10 points, where higher scores reflect greater symptom severity.
Responder rate | 1 week
  Proportion of patients with PAN-PROMISE score reduced to 6. The PAN-PROMISE score (PAtieNt-rePoRted OutcoMe scale in acute pancreatItis from an international proSpEctive cohort study) consists of a seven-item scale based on the symptoms that cause the most discomfort and concern to patients with AP. Each symptom is rated on a scale of 0 to 10 points, where higher scores reflect greater symptom severity.
Biochemical Profiles | at treatment days 3
  Mean serum IL-6 concentration at treatment days 3
Median time from AP onset to enteral nutrition resumption | an average of 1 week
  Enteral nutrition (EN) resumption refers to nutritional intake via oral or jejunal tube routes following gastrointestinal functional recovery.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The 980th Hospital of the PLA Joint Logistics Support Force (Primary Bethune International Peace Hospital of PLA), Shijiazhuang, Hebei
  - Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Department of Gastroenterology , Tangdu Hospital , Fourth Military Medical University, Xi'an, Shaanxi
  - Department of Gastroenterology, 986 Hospital of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact PI to get IPD.

REFERENCES:
- [Background] Shi X, Zhao L, Luo H, Deng H, Wang X, Ren G, Zhang L, Tao Q, Liang S, Liu N, Huang X, Zhang X, Yang X, Sun J, Qin W, Kang X, Han Y, Pan Y, Fan D. Transcutaneous Auricular Vagal Nerve Stimulation Is Effective for the Treatment of Functional Dyspepsia: A Multicenter, Randomized Controlled Study. Am J Gastroenterol. 2024 Mar 1;119(3):521-531. doi: 10.14309/ajg.0000000000002548. Epub 2023 Oct 3. PMID 37787432
- [Background] Inoue T, Abe C, Sung SS, Moscalu S, Jankowski J, Huang L, Ye H, Rosin DL, Guyenet PG, Okusa MD. Vagus nerve stimulation mediates protection from kidney ischemia-reperfusion injury through alpha7nAChR+ splenocytes. J Clin Invest. 2016 May 2;126(5):1939-52. doi: 10.1172/JCI83658. Epub 2016 Apr 18. PMID 27088805
- [Background] Morishita K, Costantini TW, Eliceiri B, Bansal V, Coimbra R. Vagal nerve stimulation modulates the dendritic cell profile in posthemorrhagic shock mesenteric lymph. J Trauma Acute Care Surg. 2014 Mar;76(3):610-7; discussion 617-8. doi: 10.1097/TA.0000000000000137. PMID 24553526
- [Background] Kelly MJ, Breathnach C, Tracey KJ, Donnelly SC. Manipulation of the inflammatory reflex as a therapeutic strategy. Cell Rep Med. 2022 Jul 19;3(7):100696. doi: 10.1016/j.xcrm.2022.100696. PMID 35858588
- [Background] Mederos MA, Reber HA, Girgis MD. Acute Pancreatitis: A Review. JAMA. 2021 Jan 26;325(4):382-390. doi: 10.1001/jama.2020.20317. PMID 33496779
- [Background] Xie J, Cai Y, Xu H, Peng Y, McArthur A. Early enteral nutrition support for patients with acute pancreatitis in the inpatient setting: a best practice implementation project. JBI Evid Implement. 2024 May 1;22(2):175-185. doi: 10.1097/XEB.0000000000000410. PMID 38415812
- [Background] Lee PJ, Papachristou GI. New insights into acute pancreatitis. Nat Rev Gastroenterol Hepatol. 2019 Aug;16(8):479-496. doi: 10.1038/s41575-019-0158-2. PMID 31138897